CLINICAL TRIAL: NCT03043612
Title: Cook Ureteral Stent Study
Brief Title: Ureteral Stent Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: 13-15
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Urolithiasis
Keywords: Ureteroscopy for urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ureteral Study Stent (Experimental): Commercially available Cook Sof-Flex® Double Pigtail Ureteral Stent that is coextruded with an alpha-blocker medication
  Interventions: Device: Cook Sof-Flex® Double Pigtail Ureteral Stent coextruded with doxazosin
- Ureteral Control Stent (Active Comparator): Commercially available Cook Sof-Flex® Double Pigtail Ureteral Stent
  Interventions: Device: Cook Sof-Flex® Double Pigtail Ureteral Stent

INTERVENTIONS:
Device: Cook Sof-Flex® Double Pigtail Ureteral Stent coextruded with doxazosin — Placement of drug-coated ureteral stent when temporary ureteral stenting is indicated following ureteroscopy for urolithiasis
  Arms: Ureteral Study Stent
Device: Cook Sof-Flex® Double Pigtail Ureteral Stent — Placement of a commercially available ureteral stent when temporary ureteral stenting is indicated following ureteroscopy for urolithiasis
  Arms: Ureteral Control Stent

SUMMARY:
The purpose of this study is to evaluate the feasibility of the Cook Ureteral Stent to reduce post-stent placement pain and urinary symptoms in patients following ureteroscopy for urolithiasis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing ureteroscopy for urolithiasis in which temporary ureteral stenting is indicated

Exclusion Criteria:

* Patient is unwilling or unable to sign and date the informed consent
* Patient is unwilling to comply with the follow-up study schedule
* Patient is pregnant, breast-feeding, or planning to become pregnant during the course of the study
* Patient is currently taking anti-cholinergic or other anti-spasm medications
* Patient is currently taking sildenafil, tadalafil, or vardenafil
* Patient has a known sensitivity to alpha-blocker medications
* Patient is currently undergoing chemotherapy or radiation therapy
* Patient has an active urinary tract infection
* Patient is in chronic renal failure, on hemodialysis, or on chronic peritoneal dialysis
* Patient requires bilateral shock wave lithotripsy, bilateral stents, or has bilateral symptomatic kidney stones
* Patient has had a ureteral stent within the past three months in either ureter
* Patient is unable to accurately detect or report bladder function or pain
* Patient has chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Patient-reported body pain score | 7-days post stent placement
  Comparing the patient-reported body pain score from the USSQ 1 survey between the two study arms

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Fai Ng, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Prince of Wales/Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No